CLINICAL TRIAL: NCT02841085
Title: Search for New Mutations Genetic Predisposing to an Increased Risk Venous Thromboembolic Disease Idiopathic. Study "FIT GENETIQUE".
Brief Title: New Genetic Mutations in Thromboembolic Venous Disease Idiopathic. Study "FIT GENETIQUE".
Acronym: Fit-Génétique
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RB 09.058 Fit Génétique
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Thromboembolic Venous Disease
Keywords: Genetic; Thrombophilia
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Genetic sample: Blood sample or saliva collection to genetic research
  Interventions: Genetic: Genetic sample

INTERVENTIONS:
Genetic: Genetic sample — Blood sample or saliva collection

SUMMARY:
Identify new genetic mutations predisposing to an increased risk of VTE by locating and / or identifying genes involved in subjects at high risk for thrombotic and in whom screening for detectable hereditary thrombophilia was negative.

DETAILED DESCRIPTION:
Venous thromboembolism desease is a public health problem justifying major primary and secondary prevention policy. When VTE occurs in the absence of risk factor clinically identifiable ( "idiopathic"), an inherited biological risk factor ( "inherited thrombophilia") is found in 30% of cases. However, in patients with idiopathic VTE, the risk of recurrent venous thromboembolism is very high, whether detectable inherited thrombophilia was found or not.

This first observation suggests that patients with idiopathic VTE and no detectable thrombophilia are likely to have an underlying unknown thrombophilia that are yet to be discovered.

This hypothesis is further supported by the results of the study "FIT" (Regional PHRC 2001, promoter CHU Brest, Investigator Main: Francis Couturaud, EA3878 Brest, France, and investigator Associate: Clive Kearon, McMaster University, Hamilton, Ontario, Canada), a cross international study evaluating the risk of VTE among the family members first degree of patients a first idiopathic VTE episode. In this large study cross-1950 family members first degree (topics study) of 372 patients with a first episode of VTE Idiopathic (propositi) were included (50% included in Brest and 50% inclusive in Canada). The main result is that the risk of VTE among family members first degree is high and similar, the proband either bearer or without a detectable hereditary thrombophilia. In other words, even in the absence of detectable hereditary thrombophilia, the risk of VTE among family members first degree is high. This study has identified the subjects in that it is likely they have an inherited thrombophilia which has not yet been discovered.

ELIGIBILITY:
Inclusion Criteria:

* Family members in the 1st, 2nd, 3rd and 4th degree (and their spouses if they have a descent) of patients (propositi) who:

  1. / have a single episode of unprovoked venous thromboembolic disease without detectable inherited and acquired thrombophilia ;
  2. / were included in the "FIT" study;
  3. / consenting that their family members 2nd, 3rd and 4th degree are approached to participate in the this study.
* Written Consent of propositi and their members in the 2nd, 3rd and 4th respective degree to participate in this study.

Exclusion Criteria:

* Presence of detectable thrombophilia in the propositi.
* Presence of hereditary thrombophilia or detectable gained at family members.
* No information may be obtained on previous venous thromboembolism among family members on 1 degree
* Everything about the study (depending on the population and members of proband Family 1st, 2nd, 3rd and 4th degree) less than 15 years.
* The family member is an adopted child

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family members in the 1st, 2nd, 3rd and 4th degree (and their spouses if they have a descent) of patients (propositi) who:
  1. / have a single episode of unprovoked venous thromboembolic disease without detectable inherited and acquired thrombophilia ;
  2. / were included in the "FIT" study;
  3. / consenting that their family members 2nd, 3rd and 4th degree are approached to participate in the this study.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2010-05-27 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Research of new genetic mutations | 1 day
  Identify new genetic mutations predisposing risk increased Thromboembolic Venous Disease by locating and / or identifying the genes involved in subjects at high risk for thrombotic and in whom screening for detectable inherited or acquired thrombophilia was negative.
  was negative.

SECONDARY OUTCOMES:
Quantify the presence of new thrombophilia hereditary risk of Thromboembolic Venous Disease | 1 day
  Quantify the importance of the presence of new thrombophilia hereditary risk of Thromboembolic Venous Disease.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France